CLINICAL TRIAL: NCT04380090
Title: Efficacy of One Dose of Laxative on Post-Operative Constipation Following Total Knee Arthroplasty
Brief Title: Post-Operative Constipation Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Kathleen Gonzalez, Interim Director of Perioperative Nursing, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-080
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Constipation
Keywords: constipation; postoperative; total knee arthroplasty
MeSH Terms: conditions — Constipation | interventions — Propylene Glycol; polyethylene glycol 3350; Dioctyl Sulfosuccinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug: Docusate Sodium (Active Comparator): Docusate sodium one pill to be taken twice a day by mouth for 28 days
  Interventions: Drug: Docusate Sodium
- Drug: Propylene Glycol (Experimental): One standard dose (17 grams) of propylene glycol by mouth on postoperative day one
  Interventions: Drug: Propylene Glycol

INTERVENTIONS:
Drug: Propylene Glycol — Patients in the propylene glycol arm will receive one standard dose of the drug on postoperative day one prior to discharge with the aim of decreasing rates of postoperative constipation for patients following single total knee replacement surgery
  Other Names: Miralax; PEG 3350
  Arms: Drug: Propylene Glycol
Drug: Docusate Sodium — Patients in the docusate sodium arm are receiving the current standard of care for prevention of postoperative constipation following single total knee replacement surgery, docusate sodium one pill twice a day by mouth for 28 days
  Other Names: Colace
  Arms: Drug: Docusate Sodium

SUMMARY:
Postoperative constipation, defined as no fully satisfying bowel movement within the first three postoperative days, is a common occurrence with some researchers estimating that between 41 and 85% of postoperative patients experience symptoms. Causes include intraoperative medications, postoperative opioid analgesics, decreased mobility, and decreased oral intake. Constipation significantly impacts quality of life following surgery. Current standard of care for preventing postoperative constipation for patients having a single total knee arthroplasty at Cleveland Clinic is discharge on postoperative day one with either a prescription to be filled for docusate sodium (brand name Colace®) 100 mg to be taken two times a day by mouth for twenty eight days or the filled prescription, plus discharge instructions on ways to avoid and treat constipation. Research results show that docusate sodium is ineffective for preventing postoperative constipation in orthopedic surgery patients, and anecdotal reports confirm this finding. The proposed study uses a 2-group non-equivalent cohort design to evaluate the effect of one standard dose (17 grams) of an over-the-counter osmotic laxative (propylene glycol (PEG 3350), brand name Miralax) by mouth prior to discharge to the current standard of care. The primary outcome measure is whether patients report of a fully satisfying, normal for them, bowel movement within the first three postoperative days. Patient reported data will be collected by phone call four to seven days following surgery. Pertinent patient characteristics will be abstracted from the electronic medical record. The sample will consist of patients over twenty years old having a single total knee arthroplasty by Drs. Stearns, Molloy, or Murray who are admitted to unit 5D at Cleveland Clinic Lutheran Hospital postoperatively. Intent to treat analysis will be performed using logistic and linear regression models, adjusting for differences between groups on patient and surgical characteristics. Based on use of a two-sided Pearson chi-square test with 80% power and significance level of 0.05, 49 patients per group are required to detect a 25% decrease in constipation rate. To account for attrition we will over sample by 50% for a total of 74 per group or 148 total participants.

ELIGIBILITY:
Inclusion Criteria:

* Admission to Cleveland Clinic Lutheran Hospital surgical unit 5D
* Single total knee replacement surgery by orthopedic surgeons Stearns, Murray, or Molloy
* Age greater than 20
* Discharge to home on postoperative day one

Exclusion Criteria:

* Known allergy to PEG 3350
* Unable to complete a follow up phone call in English
* Known renal disease, irritable bowel syndrome, or inflammatory bowel disease (Crohn's disease or ulcerative colitis)

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Gonzalez, RN, MSN, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Lutheran Hospital, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Gonzalez K, Sanchez K, Mauch K, Burchill CN, Bena JF, Morrison SL, Distelhorst KS. Efficacy of One Dose of Laxative on Postoperative Constipation Following Total Knee Arthroplasty. Orthop Nurs. 2023 Sep-Oct 01;42(5):304-309. doi: 10.1097/NOR.0000000000000971. PMID 37708528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a regional hospital within a large health system in Northeast Ohio. Recruitment began on 2/21/2020 and concluded on 7/9/2020.
Period: Overall Study
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol
Started | 76 | 78
Completed | 60 | 58
Not Completed | 16 | 20

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- Drug: Docusate Sodium: Docusate sodium one pill to was taken twice a day by mouth for 28 days
  Docusate Sodium: Patients in the docusate sodium arm received the current standard of care for prevention of postoperative constipation following single total knee replacement surgery, docusate sodium one pill twice a day by mouth for 28 days.
- Drug: Propylene Glycol: One standard dose (17 grams) of propylene glycol by mouth on postoperative day one
  Propylene Glycol: Patients in the propylene glycol arm received one standard dose of the drug on postoperative day one prior to discharge with the aim of decreasing rates of postoperative constipation for patients following single total knee replacement surgery.
- Total: Total of all reporting groups
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol | Total
Number analyzed (Participants) | 60 | 58 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (8.2) | 65.2 (9.5) | 65 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 67
  Male | 30 | 21 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 49 | 44 | 93
  Race/Ethnicity: Black/African American | 7 | 7 | 14
  Race/Ethnicity: Asian American | 1 | 1 | 2
  Race/Ethnicity: Other | 2 | 6 | 8
  Race/Ethnicity: Hispanic/Latino | 1 | 0 | 1
Saphenous Nerve Block [Count of Participants; unit: Participants]
  Yes | 59 | 57 | 116
  No | 1 | 0 | 1
  Unknown | 0 | 1 | 1
Type of anesthesia [Count of Participants; unit: Participants]
  General | 6 | 9 | 15
  Spinal | 54 | 49 | 103
Length of Surgery (minutes) [Mean (Standard Deviation); unit: Minutes] | 100.8 (20.3) | 95.7 (17.0) | 98.3 (18.8)
Quan-Charlson Comorbidity Index [Median (Inter-Quartile Range); unit: total weighted score] — The Quan Charlson Comorbidity Index (CCI) assesses comorbidity level using the number and severity of 12 pre-defined comorbid conditions. Each of the 12 items is scored between 1-6 (if present), and 0 if not present; total possible score = 28 and higher scores reflect higher comorbidity burden. The total weighted score was calculated for each subject. Median (IQR) was used in the analysis due to kurtosis.
  total weighted score | 0.00 [0.00 to 1.00] | 0.50 [0.00 to 1.00] | 0.00 [0.00 to 1.00]

OUTCOME MEASURES:

1. Primary Outcome: Bowel Movement (BM) Within 3 Days of Surgery
Description: Number of people who report normal bowel movement in the first three postoperative days following single total knee joint replacement
Time Frame: 3 days postoperative
Population: Study participants who completed the follow-up phone call
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol
Number analyzed (Participants) | 60 | 58
Participants | 29 | 32
Statistical Analysis 1: Comparison: Drug: Docusate Sodium vs Drug: Propylene Glycol; Test type: Superiority; p = 0.41, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.65 to 2.86] — OR for Propylene Glycol use (vs Docusate Sodium), adjusted for operative time and sex (female vs. male)

2. Secondary Outcome: Straining With BM
Description: For patients who had a BM within 3 days: rated 0 no straining to 10 worst straining imaginable; 3 categories developed: 0 = score of 0; 1 = score of 1-5 and 2 = score of 6-10
Time Frame: 3 days postoperative
Population: Participants who completed the follow up phone call and reported having a BM within 3 days
Measure: Number; unit: participants
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol
Number analyzed (Participants) | 29 | 32
participants
  score = 0 | 6 | 7
  score = 1 | 18 | 21
  score = 2 | 5 | 4
Statistical Analysis 1: Comparison: Drug: Docusate Sodium vs Drug: Propylene Glycol; Test type: Superiority; p = 0.66, ordinal regression model; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.28 to 2.24] — OR for Propylene Glycol use (vs Docusate Sodium), adjusted for operative time and sex (female vs. male)

3. Secondary Outcome: Pain With BM
Description: For patients who had a BM within 3 days: rated 0 no pain to 10 worst pain imaginable; 3 categories developed: 0 = score of 0; 1 = score of 1-5 and 2 = score of 6-10
Time Frame: 3 days postoperative
Population: Participants who completed the follow up phone call and reported having a BM within 3 days
Measure: Count of Participants; unit: Participants
Groups:
- Drug: Docusate Sodium: Docusate sodium one pill to be taken twice a day by mouth for 28 days Docusate Sodium: Patients in the docusate sodium arm are receiving the current standard of care for prevention of postoperative constipation following single total knee replacement surgery, docusate sodium one pill twice a day by mouth for 28 days
- Drug: Propylene Glycol: One standard dose (17 grams) of propylene glycol by mouth on postoperative day one Propylene Glycol: Patients in the propylene glycol arm will receive one standard dose of the drug on postoperative day one prior to discharge with the aim of decreasing rates of postoperative constipation for patients following single total knee replacement surgery
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol
Number analyzed (Participants) | 29 | 32
Participants
  score 0 | 19 | 19
  score 1 | 8 | 11
  score 2 | 2 | 2
Statistical Analysis 1: Comparison: Drug: Docusate Sodium vs Drug: Propylene Glycol; Test type: Superiority; p = 0.65, ordinal regression model; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.45 to 3.63] — OR for Propylene Glycol use (vs Docusate Sodium), adjusted for operative time and sex (female vs. male)

4. Other Pre Specified Outcome: Laxative Use Within 3 Days of Surgery
Description: Participant response to question: Did you take any laxatives to help you have a bowel movement in those first three days after your surgery?(yes/no) Rate of laxative use in the postoperative period was calculated for sensitivity analyses and possible adjustment of statistical models based on any group differences.
Time Frame: 3 days postoperative
Population: Study participants who completed the follow-up phone call
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol
Number analyzed (Participants) | 60 | 58
Participants | 16 | 19
Statistical Analysis 1: Comparison: Drug: Docusate Sodium vs Drug: Propylene Glycol; Test type: Equivalence — Equivalence is defined as a p-value greater or equal to 0.05 (no difference between groups); p = 0.47, Chi-squared

5. Other Pre Specified Outcome: Opioid Use Within 3 Days of Surgery
Description: Participant response to question: In the first three days following your surgery, did you take any of the opioid pain medicine prescribed by your surgeon?(yes/no) Rate of opioid use in the postoperative period was calculated for sensitivity analyses and possible adjustment of statistical models based on any group differences.
Time Frame: 3 days postoperative
Population: Study participants who completed the follow up phone call
Measure: Count of Participants; unit: Participants
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol
Number analyzed (Participants) | 60 | 58
Participants | 58 | 57
Statistical Analysis 1: Comparison: Drug: Docusate Sodium vs Drug: Propylene Glycol; Test type: Equivalence — Equivalence is defined as a p-value greater or equal to 0.05 (no difference between groups); p = 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: 7 days postoperative
Arm/Group | Drug: Docusate Sodium | Drug: Propylene Glycol
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58

LIMITATIONS AND CAVEATS:
We did not consider, in this study, the amount of opioids used by patients postoperatively. An additional limitation was that only one dose of Miralax was used in the intervention group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT04380090/Prot_SAP_000.pdf